CLINICAL TRIAL: NCT07319572
Title: Optimizing Chest Tube Removal: A Comparison of Purse-string Suture Closure and Plug Method.
Brief Title: Comparison of Chest Tube Wound Closure: Comparison Between Purse String Method and Plug Method.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Medical Sciences (Other Government)
Responsible Party: Principal Investigator, Muhammad Fahad Ali, Principal Investigator (General Surgery Resident), Pakistan Institute of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F-5-2/2024(ERCC)/PIMS
Record Dates: First submitted 2025-12-07; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Pneumothorax; Hemothorax; Chest Tube; Chest Tube Removal; Purse String; Plug Method
Keywords: Purse-string; Plug method; Chest tube; Pneumothorax; hemothorax
MeSH Terms: conditions — Pneumothorax; Hemothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Purse string group (Active Comparator): Patients in this arm will have the chest tube removal site closed using a purse-string suture technique. After chest tube removal and haemostasis, a single circumferential (purse-string) stitch is placed around the wound margin and tightened to approximate the skin edges. Skin is left approximated; additional superficial interrupted skin sutures may be applied at the investigator's discretion. Suture material: monofilament nylon or silk, per local practice. Standard sterile dressing applied. Post-procedure wound care and follow-up are identical to the comparator arm.
  Interventions: Procedure: Purse string suture closure
- Plug Method group (Experimental): After chest tube removal, the wound is swiftly plugged off with an impregnable gauze and no sutures applied. The gauze is then fixed with air tight dressing
  Interventions: Procedure: Plug method closure

INTERVENTIONS:
Procedure: Purse string suture closure — PURSE STRING METHOD OF CLOSURE: A circumferential suture is placed around the chest tube insertion site before or after tube removal. The suture is tightened like a drawstring to approximate the skin edges and close the wound. This method provides an air-tight seal but often results in a puckered, circular scar.
  PLUG METHOD OF CLOSURE: After chest tube removal, the tract is allowed to collapse naturally and is gently plugged with a small gauze piece impregnated with petroleum jelly.
  Arms: Purse string group
Procedure: Plug method closure — An impregnable gauze which is made airtight by coating it in petroleum jelly is swiftly placed over the chest wound site as the chest tube is removed and an air tight dressing done.
  Arms: Plug Method group

SUMMARY:
This prospective, comparative clinical study evaluates two techniques of chest tube wound closure-purse-string suture and the simple suture/plug method-to determine differences in cosmetic outcomes, wound complications, and overall patient satisfaction following chest tube removal. The study aims to identify the closure technique that provides optimal wound healing with fewer postoperative complications.

DETAILED DESCRIPTION:
Chest tube removal often results in small but cosmetically significant wounds. The traditional purse-string suture technique is widely used due to its presumed ability to ensure air-tight closure; however, it is frequently associated with circular or puckered scars that affect cosmetic appearance. Recently, the simple suture/plug method has been proposed as a more cosmetic alternative while maintaining adequate wound integrity.

This study prospectively enrolls patients requiring chest tube removal and allocates them to one of the two wound closure techniques. Standardized postoperative care is provided to all participants. The primary outcome is cosmetic appearance of the scar, evaluated using a validated scar assessment scale at follow-up. Secondary outcomes include wound infection, seroma or discharge, persistent air leak, wound dehiscence, time to healing, and patient satisfaction.

The findings are expected to help clinicians select the most effective and cosmetically favorable method for chest tube wound closure in routine surgical practice.

ELIGIBILITY:
Inclusion criteria :

1. All patients >18 years of age
2. Patients undergoing chest tube insertion for traumatic causes including Pneumothorax, hemothorax and hemopneumothorax.

Exclusion criteria:

1. Previous ipsilateral thoracic surgery
2. Patients with large wounds necessitating suture closure
3. Patients with bleeding disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
"Incidence of air leak after chest tube removal using purse-string suture or plug method" | 48 hours
  It is the incidence of air leak/pneumothorax after the chest tube has been removed and the wound is closed by one of the two methods of chest tube wound closure; 1) the purse string method of chest tube wound closure and 2) the plug method of chest tube wound closure.

SECONDARY OUTCOMES:
Incidence of wound infection after chest tube site closure using purse-string suture or plug method | 7 Days
  Development of surgical site infection at the chest tube removal site after closure by purse-string suture or plug method, defined according to standard surgical site infection criteria
Scar appearance score at chest tube site measured using the Vancouver Scar Scale | 1 month
  Scar quality at the chest tube removal site assessed using the Vancouver Scar Scale, which evaluates pigmentation, vascularity, pliability, and height
Patient-reported cosmetic satisfaction score after chest tube site closure measured using a Numerical Rating Scale | 1 month
  Patient-reported cosmetic satisfaction with the chest tube removal site assessed using a Numerical Rating Scale, where:
  0 = not satisfied at all
  10 = completely satisfied
  Higher scores indicate better cosmetic satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Institute of medical sciences, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Age, comorbidity, condition, locality, registration number